CLINICAL TRIAL: NCT00409630
Title: Inhaled Fluticasone Propionate: Effect on Parameters of Bone Metabolism in Patients With Mild to Moderate Asthma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided against going forward with the study.
Sponsor: University of Kansas (Other)
Collaborators: Sanofi (Industry)
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10384
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

INTERVENTIONS:
Drug: fluticasone

SUMMARY:
Subjects between the ages of 20-45 with mild to moderate asthma will be recruited. Following consent, subjects will undergo an evaluation to assure no underlying metabolic bone disease. Individuals will be treated with inhaled fluticasone low or high dose, daily for 3 months. Serum and urine biochemical markers of bone metabolism will be collected at baseline and monthly for three months. Adherence to study medication and adverse events will be collected at monthly intervals. Differences between fluticasone low and high dose treated individuals will be analyzed between groups and compared with baseline values.

DETAILED DESCRIPTION:
This study will be a prospective randomized trial. Thirty subjects with mild to moderate asthma will receive inhaled fluticasone propionate. Fifteen patients will receive low dose inhaled fluticasone 88 mcg twice daily. Fifteen patients will receive inhaled fluticasone 440 mcg twice daily. The primary outcome will be biochemical markers of bone turnover. These will include 1) serum biochemical markers of bone formation [osteocalcin, bone specific alkaline phosphatase (ALP) and procollagen I C-terminal propeptide (PICP)] and 2) markers of bone resorption, serum collagen type 1 C-Telopeptide (CTx) urinary N-telopeptide (NTx) and immunoreactive free deoxypyridinoline (iFDpd)]. Secondary endpoints will include, parathyroid hormone (PTH), Urinary Calcium/creatinine, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Before any study-specific procedure, the appropriate informed consent must be signed
* Male and premenopausal female subjects
* Age ≥ 20 years through ≤ 45 years of age
* Documented History of Mild to moderate Asthma as defined by the NHLBI guidelines:

  * Mild Intermittent - FEV1 or PEF >/= 80% predicted, PEF variability <20%.
  * Mild persistent - FEV1 or PEF >80% predicted, PEF variability, >/= 20-30%
  * Moderate persistent - FEV1 or PEF>60%-<80% predicted, PEF variability >30%
* Ambulatory status

Exclusion Criteria:

* Smoking
* Current use of inhaled glucocorticoid therapy or use within the past 3 months. Current use of leukotriene modifiers and/or inhaled bronchodilators will be allowed.
* Use of oral glucocorticoids within the past year.
* Pregnant or breast feeding.
* Last menstrual period greater than 1 year ago
* Diabetes Mellitus type 1 or 2
* Paget's Disease, osteomalacia, hyperparathyroidism, renal osteodystrophy or other metabolic bone diseases
* History of hyperthyroidism within 1 year of randomization
* AST or ALT > 2x upper limit of normal
* Serum creatinine greater than 2.0 mg/DL
* History of cancer within the previous 5 years, (exceptions: excised superficial lesions, such as basal or squamous cell carcinoma of the skin.
* The use of thiazide diuretics or anticonvulsant medications.
* Subject is currently enrolled or has received investigational drug within 30 days prior to randomization
* Use of (within 3 months of randomization) hormones, SERMS, calcitonin, PTH (Forteo)
* Use of (within 6 months of randomization) bisphosphonates, (Fosamax, Actonel, Didronel), Vitamin D 50,000 iu
* Use of (within 12 months of randomization) corticosteroids and/or inhaled steroids, anticonvulsants. Topical and intra-articular steroids are allowed except for topical steroids applied to the area where measurements of skin thickness will be made; ie.
* Use of (within 24 months of randomization) I.V. Zometa or I.V. Aredia
* Subject has any disorder that compromises the ability of the subject to give written consent and/or to comply with study procedures

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Bone markers after 3 months of fluticasone

SECONDARY OUTCOMES:
Skin thickness measured by ultrasound biomicroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Leland Graves, MD, Principal Investigator — University of Kansas Medical Center